CLINICAL TRIAL: NCT05219539
Title: Outcomes of the National Advanced Training Program for Laparoscopic Radical Gastrectomy: a Survey Based on Follow-up Questionnaire
Brief Title: Questionnaire Survey of the Advanced Training Program for Laparoscopic Radical Gastrectomy
Acronym: ATP-LRG-1
Status: Completed | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University
Other Study IDs: ATP-LRG-1
Record Dates: First submitted 2022-01-11; First posted 2022-02-02 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the outcomes of the advanced training program for laparoscopic radical gastrectomy (ATP-LRG). The research subjects are the trainees who participated in this training program.

DETAILED DESCRIPTION:
Written informed consent is not required because of the observational and anonymous nature of this study. ATP-LRG is a national training program carried out by Fujian Medical University Union Hospital. Each training lasts about 1.5 days, which includes 1) detailed technique description; 2) prevention and solving of intraoperative complications; 3) live surgery performance; 4) theory and practice of clinical research; 5) comments on trainees' videos; and 6) questions, answers and discussions. In this study, 875 trainees who participated in ATP-LRG from January 2015 to October 2020 were interviewed using electronic questionnaires. Using a repeated-measures design to examine differences in outcomes before and after participating in the training. Questionnaire Star (Changsha Ranxing Information Technology Co., Ltd), a most widely used professional online questionnaire software platform in China, was used to design and create a link to the questionnaire. The questionnaire's link was sent to each trainee via WeChat (Tencent Holdings Limited), the most commonly used social networking software in China.

ELIGIBILITY:
Inclusion Criteria:

* Participated in ATP-LRG between January 2015 and October 2020
* Have contact information

Exclusion Criteria:

* Repeated participation in ATP-LRG
* Refuse to fill out the questionnaire

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: From September 2009 to July 2021, Fujian Medical University Union Hospital have carried out 113 ATP-LRG courses, training a total of 1,447 trainees nationwide. In order to reduce recall bias, this study used an electronic questionnaire to conduct a return visit to 875 trainees who participated in the ATP-LRG for one year from January 2015 to October 2020.
Sampling Method: Non-Probability Sample
Enrollment: 1355 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Change of general surgical skills score | One year after participating in ATP-LRG
  Change of general surgical skills score = posttraining general surgical skills score - pretraining general surgical skills score. Scores were evaluated using questionares.

SECONDARY OUTCOMES:
Changes of laparoscopic gastrectomy acceptance score | One year after participating in ATP-LRG
  Changes of laparoscopic gastrectomy acceptance score = posttraining laparoscopic gastrectomy acceptance score - pretraining laparoscopic gastrectomy acceptance score. Scores were evaluated using questionares.
Changes of clinical research possibilities score | One year after participating in ATP-LRG
  Changes of clinical research possibilities score= posttraining clinical research possibilities score - pretraining clinical research possibilities score. Scores were evaluated using questionares.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China